CLINICAL TRIAL: NCT00743210
Title: Phase 1 Study of Oral L-citrulline on ADMA/L-arginine and Endothelial-dependent Vascular Function in Pregnancy.
Brief Title: Oral L-Citrulline and ADMA in Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Robert Powers, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2P01HD030367-ARG; P01HD030367-09 (NIH)
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Blood Pressure
Keywords: pregnancy; obesity; asymmetric dimethylarginine; L-arginine; L-citrulline
MeSH Terms: conditions — Obesity | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral L-citrulline, 3 grams once per day for 3 weeks.
  Interventions: Drug: L-citrulline
- 2 (Placebo Comparator): Placebo, 3 grams once per day for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-citrulline — Oral L-citrulline, 3 grams once per day for 3 weeks.
  Arms: 1
Drug: Placebo — Placebo, 3 grams once per day for 3 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if oral of L-citrulline (3 grams/day) for 3 weeks provided in mid-pregnancy to obese subjects will decrease the plasma ADMA/L-arginine ratio, lower maternal blood pressure, improve endothelial-dependent vascular function and peripheral vascular stiffness, and improve uterine artery Doppler resistance and flow.

DETAILED DESCRIPTION:
The pregnancy-specific syndrome preeclampsia is a leading cause of maternal and fetal morbidity and mortality. The underlying cause of preeclampsia is unknown, however several pre-existing maternal conditions are associated with an increased risk of preeclampsia including: diabetes, hypertension, renal dysfunction, and obesity. Among these conditions, obesity has been increasing in the population, such that 30% of the adult population in the US is now considered obese, and because of this obesity has the largest attributable risk for preeclampsia, accounting for 15 to 32% of the population attributable risk for preeclampsia. There is abundant evidence that pre-pregnancy obesity increases the risk of preeclampsia. However, it is unknown how pre-pregnancy obesity increases the risk of preeclampsia, how obesity-mediated metabolic aberrations interact with current hypotheses of the pathogenesis of preeclampsia, and why only a subset of obese women (~6-8%) develops preeclampsia. Several lines of evidence indicate that endothelial dysfunction is a central feature of the pathophysiology of preeclampsia, and endothelial dysfunction is a common endpoint of obesity. Asymmetric dimethylarginine (ADMA) is a methylated metabolite of the amino acid L-arginine and an endogenous inhibitor of nitric oxide synthase (NOS). High concentrations of ADMA contribute to endothelial dysfunction and ADMA inhibits angiogenesis and arteriogenesis, activities important in pregnancy and deficient in preeclampsia. ADMA is higher in obesity and ADMA concentrations are higher early in pregnancy among women who later develop preeclampsia. This protocol describes a randomized placebo-controlled trial of L-citrulline vs. placebo in 80 obese pregnant women from twelve to twenty weeks gestation, to determine whether L-citrulline supplementation decreases the plasma ADMA/L-arginine ratio, lowers maternal blood pressure, improves endothelial-dependent vascular function and peripheral vascular stiffness, and improvement in uterine artery Doppler resistance and flow. We will compare the data obtained from these obese pregnant women to the same measures obtained from 40 untreated lean pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy body mass index greater than or equal to 30kg/m2
* Primiparity
* Singleton pregnancy
* Gestational age at randomization between 10 and 14 weeks based on clinical information and evaluation of earliest ultrasound
* Maternal age between 14 and 40 years

Exclusion Criteria:

* chronic hypertension
* pregestational diabetes on medication (insulin, glyburide)
* major fetal anomaly or demise
* planned termination of the pregnancy
* collagen vascular disease (autoimmune disease) on medication
* renal disease
* epilepsy or other seizure disorder
* active or chronic liver disease
* heart disease
* cigarette smoker
* known illicit drug or alcohol abuse during current pregnancy
* already taking L-citrulline as a supplement (1gram/day or more)

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To evaluate blood pressure changes in response to oral L-citrulline or placebo treatment in uncomplicated obese pregnant women during the second trimester of pregnancy. | 3 weeks

SECONDARY OUTCOMES:
To evaluate the changes in plasma ADMA/L-arginine ratio, endothelial-dependent vascular function and peripheral vascular stiffness, and uterine artery Doppler resistance and flow. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Hubel, PhD, Principal Investigator — Department of Obstetrics & Gynecology and Reproductive Sciences, University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States